CLINICAL TRIAL: NCT05630261
Title: Efficacy of Internet-based Transdiagnostic Cognitive Behavioural Therapy Insomnia (CBT-I) on Comorbid Depression and Insomnia: A Pilot Randomized Controlled Trial
Brief Title: Transdiagnostic CBT-I on Comorbid Depression and Insomnia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Fiona YY Ho, Ph.D, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PSY026
Record Dates: First submitted 2022-11-20; First posted 2022-11-29 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Insomnia; Depression
Keywords: Insomnia; Depression; Cognitive behavioral therapy; Transdiagnostic; Randomized controlled trial
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-help CBT-I (Experimental): Participants assigned to the CBT-I group will receive the self-help CBT-I intervention for six weeks (i.e., participants will access the intervention every day, for 42 days).
  Interventions: Behavioral: Self-help CBT-I
- Self-help CBT-D (Active Comparator): Participants assigned to the CBT-D group will receive the self-help CBT-D intervention for six weeks (i.e., participants will access the intervention every day, for 42 days).
  Interventions: Behavioral: Self-help CBT-D

INTERVENTIONS:
Behavioral: Self-help CBT-I — The intervention will cover the following topics: (a) physiological linkage between the brain and stress, (b) sleep hygiene, (c) stimulus control, (d) sleep restriction, (e) cognitive restructuring, and (f) positive psychology. Each weekly session will be divided into 6-8 chapters. Chapters are supported by short videos and interactive games. Homework activities will be assigned after each session.
  Arms: Self-help CBT-I
Behavioral: Self-help CBT-D — The intervention will cover the following topics: (a) physiological linkage between the brain and stress, (b) emotion management, (c) cognitive restructuring, (d) behavioral activation, and (e) positive psychology. Each weekly session will be divided into 6-8 chapters. Some chapters are supported by short videos and e-worksheets. Homework activities will be assigned after each session, which include weekly record of emotions or between-session practice.
  Arms: Self-help CBT-D

SUMMARY:
This randomized control trial (RCT) aims at comparing the efficacy of self-help cognitive behavioural therapy for insomnia (CBT-I) and self-help cognitive behavioural therapy for depression (CBT-D) on comorbid depression and insomnia. It addresses the research gap of treating comorbid depression and insomnia with a transdiagnostic approach (i.e., CBT-I) rather than a disorder-specific approach (i.e., CBT-D). Insomnia is a transdiagnostic process that is common to many psychiatric disorders. It is not only a symptom for depression, but also a factor that contributes to the onset and maintenance of depression. There were limited studies comparing the efficacy of self-help CBT-I to self-help CBT-D among adults with comorbid insomnia and depression (e.g., Blom, 2015). Hence, this study will serve as one of the pioneering attempts to elucidate the role of self-help transdiagnostic insomnia therapy in reducing depressive symptoms.

Prior to all study procedures, eligible participants will be required to complete an online informed consent. Around 100 eligible participants aged between 18 and 65 with a Patient Health Questionnaire-9 score ≥ 10 indicating at least moderate level of depressive symptoms and Insomnia Severity Index (ISI) score ≥ 10 indicating clinical level of insomnia symptoms will be randomly assigned to either Internet-based CBT-I (n = 50) or Internet-based CBT-D (n = 50) in a ratio of 1:1. Eligible participants in the CBT-I group will receive the intervention "iSleepWell" via the a digital mental health platform Next Stop, Wellness! for 6 consecutive weeks, whilst the CBT-D group will receive the intervention 'LIFE FLeX' via the same platform for 6 consecutive weeks. The outcomes of interest include depressive, anxiety, and insomnia symptoms, functional impairment, quality of life, intervention credibility and acceptability at baseline (Week 0), immediate post-treatment (Week 7), and 12 weeks follow-up (Week 19) assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Hong Kong residents aged between 18 and 65;
2. Able to read and type in Chinese;
3. Have a Patient Health Questionnaire-9 (PHQ-9) score ≥ 10 indicating at least moderate level of depressive symptoms;
4. Have an Insomnia Severity Index (ISI) score ≥ 10 indicating clinical level of insomnia symptoms;
5. Have an Internet-enabled mobile device (iOS or Android operating system); and
6. Willing to provide informed consent and comply with trial protocol

Exclusion Criteria:

1. Received psychotherapy for depression and/or insomnia in the past 6 months;
2. A Patient Health Questionnaire-9 (PHQ-9) item 9 score > 2, indicating a serious level of suicidal risk (referral information to professional mental health services will be provided);
3. Any medical or neurocognitive disorder(s) that makes participation unsuitable or interferes with adherence to the proposed interventions;
4. Other untreated sleep disorders, including narcolepsy, obstructive sleep apnoea (OSA), and restless leg syndrome (RLS) / periodic leg movement disorder (PLMD) based on the SLEEP-50;
5. A change in psychotropic drugs or over-the-counter medications that target depression and/or insomnia within 2 weeks before the baseline assessment;
6. Shift work, pregnancy, or other commitments that interfere with regular sleep-wake patterns; and
7. Hospitalisation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Change in Patient Health Questionnaire | Baseline (Week 0), Immediate post-treatment (Week 7), and 12 weeks follow-up (Week 19) assessments
  The PHQ-9 is a 9-item questionnaire used for screening, diagnosing, monitoring, and measuring the severity of depression, which scores each of the nine DSM-IV criteria from "0" (not at all) to "3" (nearly every day).
Change in Insomnia Severity Index | Baseline (Week 0), Immediate post-treatment (Week 7), and 12 weeks follow-up (Week 19) assessments
  ISI is a 7-item scale designed to evaluate perceived insomnia severity. Ratings on the 5-point Likert scale are obtained on the perceived severity of sleep-onset, sleep-maintenance, early morning awakening problems, satisfaction with current sleep pattern, interference with daily functioning, noticeably of impairment attributed to the sleep problem, and level of distress caused by the sleep problem.

SECONDARY OUTCOMES:
Change in Hospital Anxiety and Depression Scale | Baseline (Week 0), Immediate post-treatment (Week 7), and 12 weeks follow-up (Week 19) assessments
  HADS is a 14-item self-rated questionnaire used for measuring the presence of anxiety and depression symptoms on a 5-point-scale.
Change in The Pittsburgh Sleep Quality Index | Baseline (Week 0), Immediate post-treatment (Week 7), and 12 weeks follow-up (Week 19) assessments
  The PSQI-19 is a 19-item questionnaire used for measuring and identifying quality of sleep. It provides a measure of global sleep quality, including sleep latency, sleep duration, habitual sleep efficiency and sleep disturbances.
Change in Sheehan Disability Scale | Baseline (Week 0), Immediate post-treatment (Week 7), and 12 weeks follow-up (Week 19) assessments
  SDS is a brief, 5-item self-report tool that assesses functional impairment in work/school, social life, and family life.
Change in Multidimensional Fatigue Inventory | Baseline (Week 0), Immediate post-treatment (Week 7), and 12 weeks follow-up (Week 19) assessments
  A 20-item self-report instrument designed to measure fatigue. Ratings on a 5-point Likert scale are obtained on the dimensions of general fatigue, physical fatigue, mental fatigue, reduced motivation and reduced activity. Scores on each subscale range from 4 to 20, with higher scores indicating greater fatigue.
Change in Short Form (Six-Dimension) Health Survey | Baseline (Week 0), Immediate post-treatment (Week 7), and 12 weeks follow-up (Week 19) assessments
  SF-6D is a preference-based single index measure of health. A six-digit number represents each SF-6D health state, each digit denotes the level of one of six SF-6D dimensions: physical functioning, role limitation, social functioning, bodily pain, mental health, and vitality. The SF-6D index, scored from 0.0 (worst health state) to 1.0 (best health state)
Change in Credibility-Expectancy Questionnaire | Baseline (Week 0) and Immediate post-intervention assessments (Week 7)
  The 6-item CEQ yielded ratings of treatment credibility, acceptability/satisfaction, and expectations for success.
Change in Treatment Acceptability/Adherence Scale | Baseline (Week 0) and Immediate post-intervention assessments (Week 7)
  TAAS is a self-reported, ten-item questionnaire that is rated by a seven-point Likert scale from 1 to 7. It aims at evaluating treatment acceptability and anticipated treatment adherence of clients in the aspects of credibility, expectancy and distress.
Demographic survey | Baseline (Week 0)
  The self-developed demographic survey will collect information including age, gender, level of education, working industry, relationship status, and location of residence, substance use, body mass index (BMI), rest-activity pattern, and social rhythms etc.

CONTACTS AND LOCATIONS:
Overall Officials: Fiona YY Ho, Ph.D, Study Chair — Chinese University of Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blom K, Jernelov S, Kraepelien M, Bergdahl MO, Jungmarker K, Ankartjarn L, Lindefors N, Kaldo V. Internet treatment addressing either insomnia or depression, for patients with both diagnoses: a randomized trial. Sleep. 2015 Feb 1;38(2):267-77. doi: 10.5665/sleep.4412. PMID 25337948